CLINICAL TRIAL: NCT04240431
Title: Symptomatic Acquired Lacrimal Passage Obstruction: Clinical Evaluation of the Level of Obstruction in Adult Patients of Upper Egypt
Brief Title: Level of Lacrimal Passage Obstruction
Status: Completed | Type: Observational
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mohamed Farag Khalil Ibrahiem, Assistant Professor, Minia University
Other Study IDs: Minia2019
Record Dates: First submitted 2020-01-21; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Lacrimal Apparatus Diseases
MeSH Terms: conditions — Lacrimal Apparatus Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Epiphora: Adult patients suffering from watering of the eye included in the study to detect level of obstruction
  Interventions: Diagnostic Test: Probing /irrigation of lacrimal passages

INTERVENTIONS:
Diagnostic Test: Probing /irrigation of lacrimal passages — Probing of the lacrimal passage was done using #00 Bowman's lacrimal probe which can reveal any narrowing (resistance) or obstruction (soft stop) of the canaliculi during its advancement from punctum towards the lacrimal sac.

SUMMARY:
Detect anatomical level of acquired lacrimal passage obstructions among patients with epiphora. They were evaluated and divided into four groups Punctal, Canalicular, Nasolacrimal duct and Mixed groups according to level of obstruction

DETAILED DESCRIPTION:
In a 3 years period adult patients with obstructive epiphora were evaluated clinically by Probing /irrigation of lacrimal passages to detect anatomical level of obstruction.

The main site of obstruction was the common canaliculus where 2/3 of patients had canalicular problems. The second common site of obstruction is nasolacrimal duct followed by the puncti.

ELIGIBILITY:
Inclusion Criteria:

* Watering of the eye
* Acquired lacrimal obstructions
* Adult patients with

Exclusion Criteria:

* No previous lacrimal surgery
* Congenital lacrimal obstructions

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were divided into four main groups according to site of narrowing or obstruction Punctal group, Canalicular group, NLD group and Mixed group who had 2 or more levels of narrowing or obstruction
Sampling Method: Non-Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-21 (Actual); Study Completion 2019-12-21 (Actual)

PRIMARY OUTCOMES:
Level of obstruction of lacrimal system | 3 years
  The level was detected either Punctal, Canalicular, Nasolacrimal duct or Mixed

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed F Ibrahiem, MD, Principal Investigator — Minia University
Locations (1):
- Faculty of Medicine, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No